CLINICAL TRIAL: NCT01749176
Title: Dulce Digital-Project Dulce 2.0 Texting Study in High Risk Latinos With Diabetes
Brief Title: Dulce Digital-Project Dulce 2.0 Texting Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: McKesson Foundation (Other); Neighborhood Healthcare (Unknown)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Dulce Digital
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes
Keywords: High risk Latino patients with diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS texting intervention (Experimental): Behavioral text messages will be sent at random times throughout the week reagarding Healthy nutrition tips, benefits of physical activity, benefits of medication adherence and requests to check blood sugar and send back results.
  Interventions: Behavioral: SMS texting intervention
- Control-Usual Care (Placebo Comparator): Participants will continue to receive their usual care in their primary care home. They will return at months 3 and 6 to conduct behavioral and laboratory assessments to compare results with the intervention group.
  Interventions: Behavioral: Control-Usual Care

INTERVENTIONS:
Behavioral: SMS texting intervention
  Arms: SMS texting intervention
Behavioral: Control-Usual Care
  Arms: Control-Usual Care

SUMMARY:
Randomized controlled trial testing the efficacy of a text messaging intervention in a low income, low health literacy group of Latino patients. Project Dulce 2.0 (PD 2.0) will address barriers to participation in health education classes, increasing adherence to treatment and medications and improving diabetes self management behaviors and skills. Two community clinic organizations that provide services to a large proportion of Latino patients with type 2 diabetes will participate to randomize 200 patients into one of 2 arms: standard diabetes management care (control) only or text messaging and standard care. Comparisons between groups will evaluate clinical, behavioral and psychosocial outcomes.

Intervention: Standard Care and Text Messaging. All participants will receive standard diabetes care provided by primary care providers at the clinic. Of the 100 that are randomized to the intervention arm will be given instructions on how the text messaging component will be addressed throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75,
* Type 2 DM,
* Enrolled at community health center,
* Latino ethnicity,
* non Project Dulce participant,
* HbA1c>/= 8%, must be able to read

Exclusion Criteria:

* Have a severe illness precluding frequent visits to the clinic,
* have a severe medical condition, poor mental function or any other reason to expect patient difficulty in complying with the requirements of the study, any history of malignancy, except subjects who have been disease-free for >10 years, or whose only malignancy has been basal or squamous cell skin carcinoma,
* patients who have a creatinine level greater than 3.5,
* any history of drug or alcohol abuse within 12 months prior to the study,
* those who are not a permanent resident in the area.
* Patients who are not willing to use a cell phone with texting capability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute
Locations (1):
- Neighborhood Health, Escondido, California, United States

REFERENCES:
- [Derived] Fortmann AL, Gallo LC, Garcia MI, Taleb M, Euyoque JA, Clark T, Skidmore J, Ruiz M, Dharkar-Surber S, Schultz J, Philis-Tsimikas A. Dulce Digital: An mHealth SMS-Based Intervention Improves Glycemic Control in Hispanics With Type 2 Diabetes. Diabetes Care. 2017 Oct;40(10):1349-1355. doi: 10.2337/dc17-0230. Epub 2017 Jun 9. PMID 28600309